CLINICAL TRIAL: NCT04723810
Title: A Study to Evaluate the Safety and Efficacy of Indocyanine Green for Intraoperative Molecular Imaging of Solid Tumors (TumorGlow™)
Brief Title: TumorGlow Intraoperative Molecular Imaging (IMI)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 844554
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Tumor, Solid
MeSH Terms: conditions — Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Patients scheduled to undergo surgical resection for the following cancers (known or suspected) that the safety and dosing/timing of indocyanine green has not been fully studied will be enrolled: glioma, breast cancer, colon cancer, rectal cancer, head and neck cancer, pulmonary metastasectomy (colorectal mets), thymoma, ovarian cancer, prostate cancer, renal cell carcinoma, thyroid cancer, parathyroid adenoma, mesothelioma, esophageal cancer, pancreas cancer, stomach cancer.
  Interventions: Drug: Indocyanine Green
- Cohort 2 (Experimental): Patients scheduled to undergo surgical resection for the following cancers (known or suspected) that the safety and dosing/timing of indocyanine green has been fully studied will be enrolled: non-small cell lung cancer, metastatic sarcoma to the lung, brain meningioma.
  Interventions: Drug: Indocyanine Green

INTERVENTIONS:
Drug: Indocyanine Green — The investigational drug is indocyanine green, single dose between 1-5 mg/kg diluted into sterile water for intravenous (IV) injection up to 5 days prior to resection surgery. The actual dose and timing from dose to imaging will be determined based on tumor type.

SUMMARY:
This is a Phase 1/2 study in patients presenting with any solid tumor and/or diseased tissue even benign nodules presumed to be resectable and at risk for recurrence on pre-operative assessment who are considered to be good surgical candidates to evaluate the safety and efficacy of the image-guided surgery using indocyanine green for intramolecular imaging of solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years of age or older.
* Patients presenting with any solid tumor and/or diseased tissue even benign nodules presumed to be resectable and at risk for recurrence on pre-operative assessment.
* Good operative candidate as determined by the treating physician and/or multidisciplinary team.
* Subject capable of giving informed consent.

Exclusion Criteria:

* Subject unable to participate in the consent process.
* Vulnerable population including pregnant women, prisoners, and children.
* History of uncontrolled hypertension (e.g., history of an ER admission for hypertensive crisis or ≥ 3 blood pressure medications)
* Patients with a self-reported history of iodide allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-01-14 (Estimated); Study Completion 2027-01-14 (Estimated)

PRIMARY OUTCOMES:
Cohort 1: Determine the safety of indocyanine green (all tumor types combined) | Up to 5 days
  Type, frequency, severity, and attribution of AEs/SAEs (all tumor types combined).
Cohort 1: Identify optimal dosing of indocyanine green before surgery, and camera combination (tumor type-specific) | Up to 5 days
  Dosing of indocyanine green, and camera combination with the highest tumor-to-background ratio (TBR) (tumor type-specific). The minimum acceptable TBR value is 2.
Cohort 1: Identify optimal timing of indocyanine green before surgery, and camera combination (tumor type-specific) | Up to 5 days
  Timing of indocyanine green, and camera combination with the highest tumor-to-background ratio (TBR) (tumor type-specific). The minimum acceptable TBR value is 2.
Cohort 2: Determine the sensitivity and specificity of indocyanine green (tumor type-specific) | Up to 5 days
  Nodule/lesion-level and subject-level sensitivity and specificity of TumorGlow (tumor type-specific).
  * Sensitivity of indocyanine green = TP/(TP+FN) = (# that fluoresce and are cancer)/(# that are cancer)
  * Specificity of indocyanine green = TN/(TN+FP) = (# that not cancer and do not fluoresce)/(# that are not cancer)
Cohort 2: Confirm the efficacy of indocyanine green used with Near Infrared (NIR) fluorescent imaging as measured by Clinically Significant Event (CSE) rate (tumor type-specific) | Up to 5 days
  Clinically Significant Event (CSE) rate (tumor type-specific). A CSE includes any of the following event:
  * One or more primary nodule (cancerous or non-cancerous) not detected under normal light and/or palpation but is detected by imaging,
  * One or more cancerous synchronous lesion not detected under normal light and/or palpation but is detected by imaging,
  * The identification of a cancer positive margin that fluoresces within (less than or equal to) 5 mm of the surgical margin.

SECONDARY OUTCOMES:
Cohort 1: Provide preliminary estimates of the sensitivity and specificity of indocyanine green (or TumorGlow) for identifying cancerous areas (tumor type-specific) | Up to 5 days
  Nodule/lesion-level and subject-level sensitivity and specificity of indocyanine green (or TumorGlow) for identifying cancerous areas (tumor type-specific).
Cohort 1: Provide preliminary estimate of the efficacy of indocyanine green for locating additional cancers and missed surgical margins as measured by CSE rate (tumor type-specific) | Up to 5 days
  Clinically Significant Event (CSE) rate (tumor type-specific).
Cohort 2: Confirm the safety of indocyanine green (all tumor types combined) | Up to 5 days
  Type, frequency, severity, and attribution of AEs/SAEs (all tumor types combined).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No